CLINICAL TRIAL: NCT02621294
Title: Measuring Protein Requirement Using the Indicator Amino Acid Oxidation Method in Healthy Young Strength and Endurance Exercise Trained Individuals
Brief Title: Measuring Protein Requirement Using Amino Acid Oxidation in Strength and Endurance Athletes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Peter Lemon, Dr., University of Western Ontario, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 004
Record Dates: First submitted 2015-11-26; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-11

CONDITIONS: Protein Requirement of Athletes
Keywords: Protein; indicator amino acid oxidation method; athletes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Measuring protein requirement (Experimental): Measuring protein requirement of athletes by feeding different amount of protein in the form of amino acid mixture and measuring their oxidation through expired CO2
  Interventions: Other: Measuring protein requirement

INTERVENTIONS:
Other: Measuring protein requirement — a repeated measures design will be used on each athlete receiving eight graded intakes of protein on separate days in the form of AA in random order ranging from 0.2 to 3.5 g/(kg/d). Three baseline samples of breath and urine will be collected at 60, 45 and 30 min before the stable isotope is given orally. During a period of 150 to 270 min. after stable isotope ingestion, 5 breath and urine samples (every 30 min) will be collected to determine an isotopic plateau in breath and urine. The rate of release of 13CO2 from the oxidation of L-[1-13C] phenylalanine (F 13CO2) in breath will be measured and a breakpoint analysis will determine total protein requirement

SUMMARY:
Our objective is to determine the dietary requirement of protein for strength and endurance exercise trained (more than 4 months training experience) individuals between 18 - 30 years of age using the indicator amino acid oxidation (IAO) method. This study will be the first to determine the required quantity of protein need per day in strength- and endurance trained young adults using the IAO method.

DETAILED DESCRIPTION:
The adequacy of the protein dietary requirement for strength (ST) and endurance (ET) exercise trained individuals has been a subject of considerable debate for many years and, at present, there is a discrepancy between those who establish dietary protein requirements for healthy adults and those issuing guidelines for athletes. Despite past nitrogen balance studies suggesting a greater protein requirement in ST and ET athletes, the Institute of Medicine (2005) recommends "no additional dietary protein for healthy adults undertaking resistance or endurance exercise". Current protein and amino acid (AA) requirement estimates for adults are based on nitrogen balance data which are considered to be flawed due to several methodological problems including the use of single linear regression for analyzing nonlinear data and an over/underestimation of nitrogen intake and excretion, respectively. To overcome these problems, the indicator amino acid oxidation technique (IAO) was developed for determination of dietary AA or protein requirements. The IAO method is based on the concept that when dietary protein is inadequate, all AA, including the indicator AA, will be oxidized. With increasing total protein intake, oxidation of the indicator AA will decrease. Once the requirement is met, there is no further change in the oxidation of the indicator AA and the inflection or 'breakpoint' is the estimated requirement. A mixed-effects change-point regression analysis to F13CO2 (label tracer oxidation in 13CO2 breath) in response to graded amounts of protein will be utilized to over come the limitations of linear regression previously used with nitrogen balance. These protein requirement measures using the IAO has not been carried out on ST or ET individuals previously so this will be the first study to do so. The results of this study will help determine the optimal protein requirement in ST and ET athletes which is important not only for athletes but also for older individuals whose loss of muscle mass has been linked to a variety of health concerns.

ELIGIBILITY:
Inclusion Criteria:

Healthy strength-trained and endurance-trained (more than 3 months training experience, at least 3x week) individuals (18-30 years old).

Exclusion Criteria:

* Unhealthy,
* sedentary individuals,
* those who are taking medication,
* those outside the age range, or
* those who have milk allergies

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
measurement of protein requirement as a response of 13C oxidation (µmol . kg-1 . h-1) of 13C-Phenylalanine to varied graded intakes of protein (g/kg/d) in form of amino acid mixture based on egg protein profile | within 8 hours of feeding period
  Oxidation of ingested L-[1-13C] phenylalanine (µmol . kg-1 . h-1) to 13CO2 (µmol . kg-1 . h-1) in response to graded intakes of protein will be measure and after determination of a plateau in oxidation curve (using change point regression analysis), break point will be defined as g/kg/d protein requirement.

SECONDARY OUTCOMES:
Measuring body composition (percent fat and fat free mass) using air displacement plethysmography (BOD POD) | 10 minutes fasted in the morning
  Participants will report fasted in the morning for the measurement of body fat and fat-free mass percent (%) using a BOD POD.
Measuring resting energy expenditure (kcal/d) using an open-circuit indirect calorimetry | 40 minutes fasted in the morning
  Resting energy expenditure (kcal/d) of all participants will be measured using an indirect calorimetry for duration of 40 min. by laying flat on a bed.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Lemon, PhD, Principal Investigator — Western University
Locations (1):
- Exercise Nutrition Research Laboratory, London, Ontario, Canada

REFERENCES:
- [Derived] Bandegan A, Courtney-Martin G, Rafii M, Pencharz PB, Lemon PWR. Indicator amino acid oxidation protein requirement estimate in endurance-trained men 24 h postexercise exceeds both the EAR and current athlete guidelines. Am J Physiol Endocrinol Metab. 2019 May 1;316(5):E741-E748. doi: 10.1152/ajpendo.00174.2018. Epub 2019 Feb 19. PMID 30779631
- [Derived] Bandegan A, Courtney-Martin G, Rafii M, Pencharz PB, Lemon PW. Indicator Amino Acid-Derived Estimate of Dietary Protein Requirement for Male Bodybuilders on a Nontraining Day Is Several-Fold Greater than the Current Recommended Dietary Allowance. J Nutr. 2017 May;147(5):850-857. doi: 10.3945/jn.116.236331. Epub 2017 Feb 8. PMID 28179492